CLINICAL TRIAL: NCT06420479
Title: The Causal Effect of Bariatric Surgery on Cardiovascular Disease and Mortality
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Conor Macdonald, Dr., Karolinska Institutet
Other Study IDs: 2024-00558-01
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Bariatric Surgery Candidate; Cardiovascular Diseases; Morality
Keywords: bariatric surgery; Cardiovascular Diseases; Mortality
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — A well-known intervention known to induce substantial weight loss

SUMMARY:
The association between weight, and cardiovascular disease and mortality is well established, however, the causal effect of weight-loss in midlife on these outcomes is less clear. Bariatric surgery results in substantial weight-loss and is an ideal candidate to study the causal effects of weight-loss. The investigators propose a project that will use causal inference and machine learning methods to answer two important questions:

1. Is bariatric surgery effective for reducing cardiovascular disease and mortality, and if so, for who?
2. Which type of bariatric surgery (gastric bypass or sleeve gastrectomy) is most effective, and for who? The investigators will use data from various Swedish registers to identify individuals with obesity who are eligible for bariatric surgery. We will then compare cardiovascular and mortality outcomes among those undergoing different types of bariatric surgery with those receiving non-surgical obesity management using causal inference methods. The investigators will use causal forests and expert knowledge to estimate indiviual treatment effects, and identify the groups of patients who benefit the most from these surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of reproductive age with a diagnosis of obesity, no prior history of cardiovascular disease or cancer, and no contraindications for surgery after 1982

Exclusion Criteria:

* Contraindications to bariatric surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of individuals eligible for bariatric surgery in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular disease | 20 year
  myocardial infarction, stroke, and death from cardiovascular causes

SECONDARY OUTCOMES:
Death from any cause | 20 year

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No